CLINICAL TRIAL: NCT02391662
Title: A Phase II Study of Nab-paclitaxel and Gemcitabine, in Elderly Patients With Previously Untreated, Metastatic Pancreatic Adenocarcinoma
Brief Title: Nab-paclitaxel and Gemcitabine, in Elderly Patients Untreated Metastatic Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asociación de Oncología Médica del Hospital de Cruces (Other)
Collaborators: Apices Soluciones S.L. (Industry); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIBABRAX; 2014-003596-27 (EudraCT Number)
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Pancreatic Carcinoma Metastatic
Keywords: Metastatic Pancreatic Adenocarcinoma; Elderly; Nab-paclitaxel; Gemcitabine
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nab-paclitaxel plus Gemcitabine (Experimental): Nab-paclitaxel 125 mg/m2 plus Gemcitabine 1000 days 1, 8 & 15 in a 28 days cycle
  Interventions: Drug: Nab-paclitaxel 125 mg/m2 weeks 1,2,3/4; Drug: Gemcitabine 1000 weeks 1,2,3/4

INTERVENTIONS:
Drug: Nab-paclitaxel 125 mg/m2 weeks 1,2,3/4 — Nab-paclitaxel 125 mg/m2 days 1,8 & 15 in a 28 days cycle
  Other Names: Nab-paclitaxel
Drug: Gemcitabine 1000 weeks 1,2,3/4 — Gemcitabine 1000 days 1,8 & 15 in a 28 days cycle
  Other Names: Gemcitabine

SUMMARY:
Cancer incidence is increasing with age and the likelihood of elderly suffering from cancer is 1:3. Although many clinical trials include elderly patients, no results for this subgroup of patients are available. Since there is no specific recommendations for treatment of elderly patients with pancreatic cancer, treatment with gemcitabine alone is the treatment of choice for these patients.

Single-agent gemcitabine is the current standard of care, but the addition of cytotoxic and targeted agents to gemcitabine has almost invariably provided no significant survival improvement.

Results obtained recently in the MPACT phase III clinical trial in patients with pancreatic cancer treated with nab-paclitaxel combined with gemcitabine have shown improvement in overall survival, but due to in this clinical trial was included patients between 27 and 88 years, it is considered necessary to conduct a specific study for patients over 70 years.

The aim of this study is to investigate whether the clinical benefit of nab-paclitaxel associated with gemcitabine can be extended to elderly patients with pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically-confirmed pancreatic adenocarcinoma
* Stage IV disease (metastatic only)
* No prior systemic therapy for their diagnosis (except in adjuvant setting > six months previously)
* ECOG performance status of 0-1
* Age >=70 years.
* Evidence of either or both of the following:

  * RECIST-defined measurable disease (lesions that can be accurately measured in at least one dimension with the longest diameter >= 20mm using conventional techniques or >= 10 mm with spiral CT scan)
  * An elevated serum CA19-9 at baseline ( >= 2X ULN)
* Female patients must be either surgically sterile or postmenopausal.
* Male patients must be surgically sterile or must agree to use a condom during sex with women who may become pregnant while receiving the study drug and for 6 months after receiving the last dose.
* Adequate bone marrow function:

  * ANC >= 1500/uL
  * platelet count >= 100,000/uL
  * hemoglobin >= 9.0 g/dL
* Adequate hepatic function:

  * Total bilirubin <= 1.5 X ULN
  * AST (SGOT) <= 2.5 X ULN
  * ALT (SGPT) <= 2.5 X ULN
* Adequate renal function as determined by either:

  * Serum creatinine <= 1.5 X ULN
  * Calculated or measured creatinine clearance >= 40 mL/min (for calculated creatinine clearance, Cockroft-Gault equation will be used).
* Ability to understand the nature of this study protocol and give written informed consent
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Any prior systemic or investigational therapy for metastatic pancreatic cancer.
* Inability to comply with study and/or follow-up procedures.
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that, in the opinion of the investigator, renders the subject at high risk from treatment complications or might affect the interpretation of the results of the study.
* Presence of central nervous system or brain metastases.
* Life expectancy < 12 weeks.
* Pregnancy (positive pregnancy test) or lactation.
* Prior malignancy except for adequately treated basal cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other form of cancer from which the patient has been disease-free for 5 years.
* Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months.
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.
* Known, existing uncontrolled coagulopathy.
* Pre-existing sensory neuropathy > grade 1.
* Major surgery within 4 weeks of the start of study treatment, without complete recovery.
* Concurrent/pre-existing use of anticoagulant treatment.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-06-23 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment through 3-months deterioration free rate | Up to 3 months
  The general deterioration of the patient is assessed with the EORTC-QLQ-C30 scale. t will be considered definitive deterioration a decrease of at least 10 points from baseline. We will evaluate the rate of patients free of definitive deterioration at 3 months.

SECONDARY OUTCOMES:
Evaluate safety profile of gemcitabine and nab-paclitaxel, measured by Number of events per patient according to NCI-CTC-AE criteria | Up to 6 months
  Number of events per patient according to NCI-CTC-AE criteria
Time to tumor progression | Up to 8 months
  Time from patient inclusion to disease progression according RECIST criteria
Overall survival | Up to 12 months
  Time from patient inclusion to death
Objective radiographic response (ORR) | Up to 6 months
  Response rate will be evaluated according RECIST criteria
CA 19.9 biomarker response | Up to 6 months
  CA 19.9 biomarker response will be considered a decrease of at least 50% compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo López Vivanco, MD, Study Chair — Hospital de Cruces
Locations (21):
- Spain (21):
  - Hospital General de Granollers, Granollers, Barcelona
  - Centre Hospitalari de Manresa, Manresa, Barcelona
  - Hospital Universitario de Cruces, Barakaldo, Gipuzkoa
  - Hospital Clinico Universitario Virgen de La Arrixaca, El Palmar, Murcia
  - Hospital Xeral de Vigo, Vigo, Pontevedra
  - Complejo Hospitalario Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Infanta Cristina, Badajoz
  - Hospital Universitario Vall D'Hebron, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Ico Girona, Girona
  - Complejo Hospitalario de Jaén, Jaén
  - C. Hospitalario Universitario Insularmaterno-Infantil, Las Palmas de Gran Canaria
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Hm Sanchinarro, Madrid
  - Hospital Quirón Madrid, Madrid
  - Complexo Hospitalario Universitario de Ourense, Ourense
  - Complejo Hospitalario Regional Virgen Macarena, Seville
  - Hospital Virgen Del Rocio, Seville